CLINICAL TRIAL: NCT00836537
Title: A Relative Bioavailability Study of 40 mg Benazepril Hydrochloride Tablets Under Non-Fasting Conditions
Brief Title: Benazepril HCl 40 mg Tablets, Fed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R01-050
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — benazepril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Benazepril HCl 40 mg Tablets
- 2 (Active Comparator)
  Interventions: Drug: Lotensin® 40 mg Tablets

INTERVENTIONS:
Drug: Benazepril HCl 40 mg Tablets — 1 x 40 mg, single-dose fed
  Arms: 1
Drug: Lotensin® 40 mg Tablets — 1 x 40 mg, single-dose fed
  Arms: 2

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 40 mg Benazepril Hydrochloride Tablets by TEVA Pharmaceuticals Industries, Ltd. with that of 40 mg LOTENSIN® Tablets by Novartis Pharmaceuticals following a single oral dose (1 x 40 mg) in healthy adult volunteers under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers for selected for this study will be healthy men or women 19 years of age or older at the time of dosing. The weight range will not exceed ±20% for height and body frame as per Desirable Weights for Men - 1983 Metropolitan height and Weight Table or as per Desirable Weights for Women - 1983 Metropolitan Height and Weight Table. Subjects must have a minimum weight of at least 110 pounds.
* Screening procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.

Screening will include general observations, physical examination, demographics, medical and medication history, a 12-lead electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.

* The screening clinical laboratory procedures will include:

  1. Hematology: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count;
  2. Clinical Chemistry: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase;
  3. HIV antibody, hepatitis B surface antigen, and hepatitis C antibody screens;
  4. Urinalysis: by dipstick; full microscopic examination if dipstick positive; and
  5. Urine Drug Screen: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine.
  6. Serum Pregnancy Screen (female volunteers only)
* If female and:

  1. of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, sponge, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
  2. is postmenopausal for at least 1 year; or
  3. is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse in the past 24 months.
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined bt the medical investigator).
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Volunteers demonstrating a positive hepatitis B surface antigen screen, hepatitis C antibody screen or a reactive HIV antibody screen.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Female volunteers demonstrating a positive pregnancy screen.
* Female volunteers who are currently breastfeeding.
* Volunteers with a history of allergic response(s) to benazepril hydrochloride or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the medical investigator).
* Volunteers who currently use tobacco products. Three months abstinence is required.
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to Period I dosing.
* Volunteers who report donating greater than 150 mL of blood within 30 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weks after completing the study.
* Volunteers who report receiving any investigational drug within 30 days prior to period I dosing.
* Volunteers who report taking any prescription medication in the 14 days prior to Period I dosing and no OTC medications within 7 days prior to Period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-03; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax for Benazepril | Blood samples collected over 96 hour period
Bioequivalence based on AUC0-inf for Benazepril | Blood samples collected over 96 hour period
Bioequivalence based on AUC0-t | Blood samples collected over 96 hour period

SECONDARY OUTCOMES:
Cmax results for Benazeprilat | Blood samples collected over 96 hour period
AUC0-inf results for Benazeprilat | Blood samples collected over 96 hour period
AUC0-t results for Benazeprilat | Blood samples collected over 96 hour period

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson, Pharm. D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States